CLINICAL TRIAL: NCT00653965
Title: A 6-Week, Randomized, Open-Label, Comparative Study to Evaluate the Efficacy and Safety of Rosuvastatin and Atorvastatin in the Treatment of Hypercholesterolaemia in Hispanic Subjects.
Brief Title: Treatment of Hypercholesterolaemia in Hispanic Subjects (STARSHIP)
Acronym: STARSHIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522US/0007; D3560L00027
Record Dates: First submitted 2008-03-26; First posted 2008-04-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia; Dyslipidaemia
Keywords: Cholesterol; low density lipoproteins; dyslipidaemia; Rosuvastatin; Crestor; Atorvastatin; Lipitor; Hispanic
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of 6 weeks of treatment with Rosuvastatin with 6 weeks of treatment with Atorvastatin in Hispanic subjects with hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Fasting low density lipoprotein & triglyceride levels as defined by the protocol.
* Self described Hispanic race
* Subjects with coronary heart disease or at high risk of coronary heart disease.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Blood lipid levels above the limits defined in the protocol.
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2003-05; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Low density lipoproteins cholesterol levels | 6 weeks

SECONDARY OUTCOMES:
Other blood lipid level changes | 6 weeks
Safety: adverse events & abnormal laboratory markers | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Haffner, MD, Principal Investigator — San Antonio, USA; Russell Esterline, Study Director — AstraZeneca